CLINICAL TRIAL: NCT01898104
Title: Phase 1/2 Study of Valproic Acid and Short-course Radiotherapy Plus Capecitabine as preoperatIve Treatment in Low-moderate Risk Rectal Cancer
Brief Title: Preoperative Valproic Acid and Radiation Therapy for Rectal Cancer
Acronym: V-shoRT-R3
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V-shoRT-R3; 2012-002831-28 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer
Keywords: rectal; low risk; moderate risk
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Valproic Acid; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SCRT (Active Comparator): short course radiotherapy (SCRT) alone 25 Gy in 5 fractions over one week.
  Interventions: Radiation: preoperative radiation therapy
- V-SCRT (Active Comparator): Valproic acid (V) + short course radiotherapy
  Interventions: Radiation: preoperative radiation therapy; Drug: Valproic Acid
- C-SCRT (Active Comparator): capecitabine (C) + short course radiotherapy
  Interventions: Radiation: preoperative radiation therapy; Drug: Capecitabine
- VC-SCRT (Active Comparator): valproic acid + capecitabine + short course radiotherapy
  Interventions: Radiation: preoperative radiation therapy; Drug: Valproic Acid; Drug: Capecitabine

INTERVENTIONS:
Radiation: preoperative radiation therapy — 25 Gy in 5 fractions over 1 week
Drug: Valproic Acid
  Arms: V-SCRT; VC-SCRT
Drug: Capecitabine
  Arms: C-SCRT; VC-SCRT

SUMMARY:
The purpose of this study is to first determine the maximum tolerated dose of capecitabine given alone or in combination with valproic acid during preoperative short-course radiotherapy (Phase 1). The next part of the study (Phase 2)will explore whether the addition of valproic acid or the addition of capecitabine to short-course radiotherapy, before optimal radical surgery might increase the pathologic complete tumor regression rate in patients with low-moderate risk rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

• Patients with histologically confirmed diagnosis of adenocarcinoma of rectum falling into one of the following categories: T2N0 located at <2 cm from anal verge T2N1 or T3N0-N1, located at >5 cm and <12 cm from anal verge and infiltration of perirectal fat up to a distance of 1 mm from mesorectal fascia (MRF) evaluated by MRI.

* Age ≥18 and ≤ 70
* ECOG Performance Status ≤1
* Effective contraception for both male and female patients if the risk of conception exist
* Signed written informed consent

Exclusion Criteria:

* Any previous treatment for rectal cancer
* Previous pelvic radiotherapy
* Presence of metastatic disease
* Recurrent rectal tumor
* Patient with Familial Adenomatosis Polyposis (FAP) or Hereditary Non-Polyposis Colorectal Cancer (HNPCC)
* History of inflammatory bowel disease or active disease
* Any concurrent malignancy except for adequately treated basocellular carcinoma of the skin or in situ carcinoma of cervix uteri. Patients with a previous malignancy but without evidence of disease for 5 years will be allowed to enter the trial.
* Neutrophils < 2000/mm3 or platelets < 100.000/ mm3 or haemoglobin <9 gr/dl.
* Creatinine levels indicating renal clearance of <50 ml/min
* GOT and/or GPT > 2.5 time the UNL and/or bilirubin >1.5 time the upper-normal limits (UNL)
* Significant cardiovascular comorbidity (e.g. myocardial infarction, superior vena cava [SVC] syndrome, patients with an ejection fraction of <50%) or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia.
* Patients with long QT-syndrome or QTc interval duration > 480 msec or concomitant medication with drugs prolonging QTc (see list in the appendix)
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* HIV positive patients
* Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
* Known or suspected hypersensitivity to any of the study drugs.
* Patient who have had prior treatment with an HDAC inhibitor and patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid.
* Concurrent uncontrolled medical conditions that might contraindicate study drugs.
* Major surgical procedure, within 28 days prior to study treatment start.
* Pregnant or lactating women.
* Women of childbearing potential with either a positive or no pregnancy test at baseline (NB. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2012-05; Primary Completion 2023-11 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose of capecitabine, given alone or in combination with valproic acid | up to 3 weeks
  Phase 1 primary objective
number of patients with complete pathological tumor regression | 8 weeks
  evaluated at definitive surgery, planned 8 weeks after the end of radiotherapy, in all the study arms of Phase 2

SECONDARY OUTCOMES:
overall survival | 1 year
number of patients alive with disease progression | one year
number of patients with pathologic complete response | 2 months
changes in quality of life from baseline | up to 3 months

OTHER OUTCOMES:
evaluation of predictive factors | 2 months
  description of predictive role of early tumor metabolic changes measured by PET scan
predictive and prognostic factors of tumor and circulating cells | 2 months
  descriptive exploratory analyses

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Avallone, M.D., Principal Investigator — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Italy

REFERENCES:
- [Derived] Avallone A, Piccirillo MC, Delrio P, Pecori B, Di Gennaro E, Aloj L, Tatangelo F, D'Angelo V, Granata C, Cavalcanti E, Maurea N, Maiolino P, Bianco F, Montano M, Silvestro L, Terranova Barberio M, Roca MS, Di Maio M, Marone P, Botti G, Petrillo A, Daniele G, Lastoria S, Iaffaioli VR, Romano G, Caraco C, Muto P, Gallo C, Perrone F, Budillon A. Phase 1/2 study of valproic acid and short-course radiotherapy plus capecitabine as preoperative treatment in low-moderate risk rectal cancer-V-shoRT-R3 (Valproic acid--short Radiotherapy--rectum 3rd trial). BMC Cancer. 2014 Nov 24;14:875. doi: 10.1186/1471-2407-14-875. PMID 25421252